CLINICAL TRIAL: NCT04282512
Title: Evaluation of the Effect of Daily Consumption of Sodium Bicarbonate Water for 15 Days on Blood Pressure in Normotensive Subjects
Brief Title: Evaluation of the Effect of Sodium Bicarbonate Water on Blood Pressure in Normotensive Subjects
Acronym: ROX_TENSIO18
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: My Goodlife SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MGL-003
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Blood Pressure
Keywords: Nutrition; Blood pressure; Sodium bicarbonate

STUDY DESIGN:
Intervention Model Description: Group A subjects: first 15-day period drinking a sodium bicarbonate-rich mineral water Group B subjects: first 15-day period drinking tap water Washout period of 15 days Group A subjects: last 15-day period drinking tap water Group B subjects: last 15-day period drinking a Sodium bicarbonate-rich mineral water
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A : sodium bicarbonate-rich mineral water and tap water (Experimental): First 15-days period with daily intake of 1.5l of sodium bicarbonate-rich mineral water.
  15-days washout period Last 15-days period with daily intake of 1.5l of tap water.
  Interventions: Other: Sodium bicarbonate-rich mineral water
- Group B : tap water and sodium bicarbonate-rich mineral water (Experimental): First 15-days period with daily intake of 1.5l of tap water. 15-days washout period Last 15-days period with daily intake of 1.5l of sodium bicarbonate-rich mineral water.
  Interventions: Other: Sodium bicarbonate-rich mineral water

INTERVENTIONS:
Other: Sodium bicarbonate-rich mineral water — St-Yorre, a sodium bicarbonate-rich mineral water, is a commercial mineral water that contains 4368 mg/l sodium bicarbonate. The study intends to evaluate the effect on blood pressure of the sodium bicarbonate intake due to this mineral water consumption.
  Other Names: St-Yorre mineral water

SUMMARY:
ROX_TENSIO18 is a randomised cross-over trial and the main objective is to evaluate the effect of daily consumption of sodium bicarbonate water for 15 days on blood pressure.

Secondary objective are:

* Evaluation of the effect of daily consumption of sodium bicarbonate water on total salt intake
* Evaluation on blood pressure of the usual food groups that are the strongest contributors of salt intake.

DETAILED DESCRIPTION:
Volunteers are normotensive subjects divided into two equivalent groups. Group A subjects will begin their first 15-day period with the consumption of St-Yorre mineral water.

Group B will begin the first 15-day period by drinking tap water. After a washout period of 15 days, each group alternates with a new period of 15 days of water consumption monitoring: tap water for group A and mineral water St-Yorre for group B.

For each period salt intake and blood pressure are measured.Three-day food records are also performed for both 15-days periods.

ELIGIBILITY:
Inclusion Criteria:

* Normal blood pressure between 90/60 and 140/90 mm Hg
* Usually drinks tap water;
* Knowing read and write French routinely,
* Possessing an internet connection at home,
* Possessing and knowing how to use a computer or tablet,
* Affiliated with a social security scheme
* Not Trust
* Having signed the informed consent letter

Exclusion Criteria:

* Pregnant or lactating woman
* BMI greater than 35 kg / m²
* Heart failure
* History of cardiovascular disease
* Hypertension treated or untreated
* Renal failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline mean number of systolic and diastolic blood pressure at 15 days | Day 1 to Day 3 - Day 13 to Day 15- Day 31 to Day 33 - Day 43 to Day 45
  The primary endpoint is the difference between mean number of blood pressure of the volunteers drinking sodium bicarbonated-rich water during 15 days and the mean number of volunteers drinking tap water during 15 days.

SECONDARY OUTCOMES:
Sodium intake | Day 1 to Day 15 - Day 31 to Day 45
  The sodium intake per day is assessed using two three-day food records and the ExSel test.

CONTACTS AND LOCATIONS:
Overall Officials: Saïd Bekka, MD, PhD, Principal Investigator — INSTITUT DE DIABÉTOLOGIE ET NUTRITION DU CENTRE
Locations (1):
- Institut de Diabétologie Et Nutrition Du Centre, Mainvilliers, France

IPD SHARING:
Plan to Share IPD: No